CLINICAL TRIAL: NCT02994693
Title: Natural History of Barrett's Esophagus Using Tethered Capsule Endomicroscopy
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator - MD, PhD, FACC, FCAP, FNAI, Massachusetts General Hospital
Other Study IDs: 2016-P000919; 5R01CA184102-02 (NIH)
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Barrett Esophagus; Barretts Esophagus With Dysplasia
Keywords: Barrett's Esophagus; Natural History; Device; OCT; Capsule; Tethered Capsule Endomicroscopy
MeSH Terms: conditions — Barrett Esophagus | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- OFDI capsule imaging: Participants will swallow the OFDI capsule and imaging will be acquired using the OFDI imaging system.
  Interventions: Device: OFDI capsule imaging

INTERVENTIONS:
Device: OFDI capsule imaging — Imaging of Barrett's esophagus (BE) using OFDI capsule imaging

SUMMARY:
The goal of this research is to determine the natural history of Barrett's esophagus (BE) using tethered capsule endomicroscopy (TCE) in participants undergoing surveillance endoscopy.

DETAILED DESCRIPTION:
The MGH will be the first site in the multi-center study to begin enrolling. At the MGH 100 participants with a previous diagnosis of Barrett's Esophagus (BE) will be enrolled.

Each subject will undergo a minimum of 2 esophagogastroduodenoscopies (EGD), one around the time of inclusion into the study and one at the end of the study, and 4 TCE imaging sessions (baseline, 1-year, 2-years and at the end of the 3-years follow-up). If it is determined by the treating physician that additional EGDs are needed, for extended follow-up or treatment, capsule imaging will be performed whenever possible.

Participants will have received written information prior to the day of the capsule procedure and participants will have another chance to discuss the procedure with the study coordinator and clinical study staff during the consent process prior to the capsule procedure. Participation in this study is completely voluntary, and the participant can stop the procedure at any time.

For each of the imaged participants, inclusion criteria and clinical characteristics such as age, sex, body mass index (BMI), current medication regimen, smoking history and GI related history will be recorded in the clinical form.

Participants will be seated and asked to sip water to facilitate swallowing the capsule.

The device will be operated by experienced study staff trained in the procedure such as a registered nurse or one of the endoscopist co-investigators in this study. Emergency phone and/or pager contact of the collaborating GI clinician(s) will be provided. They will also be accessible during the procedure if any problems are encountered that require their expertise.

Imaging will be performed in the same manner as in our other current IRB approved tethered capsule endomicroscopy studies. The capsule position will be controlled manually via the tether outside of the participant's mouth by the catheter operator. Recorded real-time cross-sectional images displayed on the monitor and distance marks on the tether will be used for confirmation of capsule position in the esophagus. Images will be viewed in real time to determine when the capsule has reached the stomach. The resistance of the tether can also give information of the cardia position. Once in the stomach, the capsule will be gradually pulled back up through the esophagus to the mouth, also while imaging. The capsule may be repositioned for imaging up to 4 times up and 4 times down the esophagus. The participant may be asked to swallow a different size capsule (ranging from 5-12.8 mm in diameter and 20-30 cm in length) to obtain the best distal esophageal images. It is expected that the maximum experimental time including swallowing the capsule, the imaging procedure, and removal of the capsule will take approximately 10 minutes in total.

ELIGIBILITY:
Inclusion Criteria:

* Participants with known BE without high grade dysplasia, intramucosal adenocarcinoma or esophageal adenocarcinoma, confirmed by endoscopic biopsy,
* Participants over the age of 18
* Participants who are capable of giving informed consent
* Participants who had or will have a standard of care EGD within 9 to 15 months
* Participants must have no solid food for at least 4 hours prior to the procedure, and only clear liquids for 2 hours prior to the procedure.

Exclusion Criteria:

* Participants with prior endoscopic ablation or resection treatment of BE
* Participants with esophageal fistula and/or esophageal strictures with a luminal stricture diameter that is smaller than the diameter of the capsule
* Participants with the inability to swallow capsules.
* Pregnancy, according to participant information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with known BE without high grade dysplasia, intramucosal adenocarcinoma or esophageal adenocarcinoma, confirmed by endoscopic biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Longitudinal assessment of the Natural History of Barrett's Esophagus Using Tethered Capsule Endomicroscopy | Approximate 25 minutes visit (10 min image acquisition)
  An investigator will assess the quality of the recorded images and movies obtained with each exam after imaging has been completed. They will assess how the images change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong J, Grant C, Vuong B, Nishioka N, Gao AH, Beatty M, Baldwin G, Baillargeon A, Bablouzian A, Grahmann P, Bhat N, Ryan E, Barrios A, Giddings S, Ford T, Beaulieu-Ouellet E, Hosseiny SH, Lerman I, Trasischker W, Reddy R, Singh K, Gora M, Hyun D, Queneherve L, Wallace M, Wolfsen H, Sharma P, Wang KK, Leggett CL, Poneros J, Abrams JA, Lightdale C, Leeds S, Rosenberg M, Tearney GJ. Feasibility and Safety of Tethered Capsule Endomicroscopy in Patients With Barrett's Esophagus in a Multi-Center Study. Clin Gastroenterol Hepatol. 2022 Apr;20(4):756-765.e3. doi: 10.1016/j.cgh.2021.02.008. Epub 2021 Feb 4. PMID 33549871